CLINICAL TRIAL: NCT05538442
Title: Kinetics of the Determinants of Performance During an Ultra-trail
Brief Title: Trail Sciences Clecy: Markers of Performances
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2021-A01765-36
Record Dates: First submitted 2022-01-31; First posted 2022-09-13 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-01

CONDITIONS: Sports Injury
Keywords: Ultra trail; effort physiology; thermoregulation; tiredness; sleep deprivation; biology
MeSH Terms: conditions — Athletic Injuries; Fatigue; Sleep Deprivation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- group (Other): Healthy trailer
  Interventions: Other: Physiological recordings

INTERVENTIONS:
Other: Physiological recordings — Physiological, cognitive, biological measurments

SUMMARY:
The Scientific Trail Protocol of Clécy - Suisse Normande (TCS) is exploratory study including several specific protocols, on a real event of 156 km on hilly terrain (6000 m of difference in level), allowing to evaluate the constraints and immediate (6000 m of difference in altitude), allowing to evaluate the constraints and the immediate physiological adaptations under race conditions.

The evaluations will be performed by collecting biological and neurobiological variables before, during and after the race (inflammation, hydro-electrolytic, cardiac, renal and muscular balance), physiological parameters whose thermoregulatory processes (core temperature, skin temperature, hydration), neuromuscular fatigue, cognitive performances (motivation, attention, emotion) and sleep changes (before, during and after the race).

DETAILED DESCRIPTION:
Running has deep evolutionary roots in human history. The ability and the ability and propensity to run long distances would have appeared about 2 million years ago when humans were hunting to exhaustion in order to feed themselves with meaty foods. Today, these exceptional endurance abilities are the modern manifestation of a unique human trait that helps make humans what they are.

For 20 years, the popularity of ultra-endurance disciplines (effort whose duration is greater than 6 hours) is exponential. Ultra-trail in particular has not escaped this popular worldwide craze. At the same time, the scientific community, particularly the medical community, is beginning to take an interest in this discipline. It is important to It is important to understand how a human organism is able to produce an effort of several tens of hours hours continuously. It is necessary to measure the short, medium and long term repercussions on the health of It is necessary to measure the short, medium and long term repercussions on the health of ultra-trail to ensure its development and its practice in complete safety, in a society that is becoming more and more sedentary.

The lack of data found in the literature on these issues is essentially related to the the difficulty of setting up scientific protocols during events, associated with the preponderant place of the trail discipline, on which the project in Clécy,Normandy is originated.

A consortium composed of several local research teams (Normandy Caen University Hospital), national and international research teams, propose to set up a common protocol to better explore and understand the time course of the psychophysiological mechanisms that contribute to performance during an ultra trail. For this purpose, measurements will be taken before, during and after the Ultra Trail (156 km) in 60 voluntary and experienced runners. This scientific study, so complete with a dedicated race, is the first of its type in ultra-trail.

This experimental study will include 60 subjects, men and women, experienced in ultra trail running events and with no contraindications to the practice of this discipline.

This experimental group will participate in a 156 km / 6000mD+ race (between 24 and 60 hours of running) and will take measurements at each lap (every 26 km). Hypothesis tested: The aim of this work is to evaluate the time course of parameters contributing to the performance/skills during a run of 156 km with a positive elevation difference of 6000 m.

ELIGIBILITY:
Inclusion Criteria:

Medical certificate of no contraindication to the practice of the ultra trail of less than one year and having no abnormalities in the ECG nor in the cardiac echography realized in the 2 months preceding the race.

* Runners voluntarily participating in the Trail Scientifique de Clécy (156 Km / 6000D+)
* Experienced runners who have already completed 2 ultra trail races (+/- 160km), at least one of them in the last 24 months. The subjects will have to justify their event and their ranking.
* Be affiliated to a social security system or be a beneficiary of such a system Plan
* Free and informed information given to the participant
* French language spoken and read
* Healthy volunteers from 25 years old to 60 years old.
* Ability to give written consent to participate in the study.
* Usual place of living: Greenwich meridian (GMT) ± 2 hours
* Be equipped with a cardio-gps watch (Suunto, Polar, Garmin, Coros) and a Android smartphone
* Subjects who have not run a trail of more than 80 km in the 3 weeks preceding the protocol
* All participants will have to present a health pass under the legislation in force on November 11

Exclusion Criteria:

* Subjects with a medical history (pulmonary pathology, cardiac pathology, hypertension) or with known inflammatory, renal, cardiac or neurological disease.
* History of joint surgery of the ankle (e.g. arthrodesis) or foot.
* Pathology / trauma of the lower limbs
* Joint stiffness corresponding to amplitudes of less than 15° of dorsal flexion (flexion) and 35° of plantar flexion (extension)
* Major sensory disorders in the foot (loss of sensitivity).
* Central and/or peripheral neurological pathology
* Swallowing disorder.
* Chronic transit disorder (UC, Crohn's disease, digestive cancer...) Recent muscular and orthopedic injuries limiting running (less than 15 days)
* Participants who have experienced a time difference of more than 2 hours in the month preceding the event (jet lag)
* Subject having run an ultra-trail (160 Km) after the period of September 2 2021
* Pregnant or breastfeeding woman
* Minor subject
* Inclusion of the subject in another biomedical research protocol during the present study
* Patient under guardianship or curatorship
* Refusal of participation, impossibility to access or read the information letter
* MRI scheduled within 48 hours after the race
* Runner under medical treatment.
* Physical or mental inability to perform the isokinetic test
* Absence of a valid health pass

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-11-09 (Actual); Primary Completion 2021-11-14 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Core body temperature 1 changes from baseline | continuous monitoring from Day 1 before (baseline) to Day 2 after the ultra-trail
  Continuous monitoring of Measurment of body core temperature with e-celcius device for circadien rythm measurments.
Biomechanical properties1 | Comparison at the end of the race from baseline before race
  To study the variation of passive myotendinous mechanical properties of the suro-spinal complex by elastography techniques.
  - Maximum tension interpreted by peak torque at 10° of dorsal flexion (peak torque: PT in Nm)
Biomechanical properties2 | Comparison at the end of the race from baseline before race
  To study the variation of passive myotendinous mechanical properties of the suro-spinal complex by elastography techniques.
  - Stiffness interpreted by the Tension/Length ratio: ΔPT/ΔL at 0-10° of extension
Biomechanical properties3 | Comparison at the end of the race from baseline before race
  To study the variation of passive myotendinous mechanical properties of the suro-spinal complex by elastography techniques.
  - Elastic potential energy (W) interpreted by the area under the PT-L curve 0-10° of extension
Spatial cognition evaluations from baseline | Comparison at the end of the race from baseline before race
  Evaluation of spatial orientation through virtual reality orientation test (XMaze, VRMaze software)
Balance evaluations 1 from baseline | Comparison at the end of the race from baseline before race
  Evaluation of balance ability through posture measurments antero-posterior and lateral sway during eye open and closed condition
Balance evaluations 2 from baseline | Comparison at the end of the race from baseline before race
  Evaluation of balance ability through posture measurments through the stability score during eye open and closed condition
Sleep scoring changes from baseline | Comparison at the end of the race from baseline before race
  Sleep recordings with the somfit EEG device and quantification of wake, NREM and REM states duration.
Sleep scoring through actimetry | Comparison at the end of the race from baseline before race
  Continuous actimetric monitoring through a motion watch
Sleep scoring through heart frequency | Comparison at the end of the race from baseline before race
  Continuous monitoring of heart rate with a physiological suit
Cardio-vascular evaluations changes from baseline | Comparison at the end of the race from baseline before race
  Estimation of acute variations of left ventricular relaxation in echocardiography echocardiography by measuring left proto-diastolic intraventricular pressure gradients
cognitive processes 1 changes from baseline | Comparison at the end of the race from baseline before race
  Determine how cognitive performance (decision making, alertness) is altered by the test and discriminate the effect of exercise and sleep disturbance.
  Test to measure attention: PVT (Vigilance, 3 min)
cognitive processes 2 changes from baseline | Comparison at the end of the race from baseline before race
  Determine how cognitive performance (decision making, alertness) is altered by the test and discriminate the effect of exercise and sleep disturbance.
  DSST cognitive test (Complex Deciphering and Visual Tracking, 90 seconds)
cognitive processes 3 changes from baseline | Comparison at the end of the race from baseline before race
  Determine how cognitive performance (decision making, alertness) is altered by the test and discriminate the effect of exercise and sleep disturbance.
  BART Cognitive Test (Risk Decision Making, 3 min)
shoes related biomechanic 1 changes from baseline | Comparison at the end of the race from baseline before race
  To study the relationship between the pair of shoes worn and the morphological, biomechanical and sensory characteristics of the ultra-endurance runner- Measurement of foot dimensions (scanner)
  - Collection of stated footwear preferences (questionnaire)
shoes related biomechanic 2a changes from baseline | Comparison at the end of the race from baseline before race
  To study the relationship between the pair of shoes worn and the morphological, biomechanical and sensory characteristics of the ultra-endurance runner- Measurement of foot dimensions (scanner)
  - Measurement of biomechanics (foot placement technique)
shoes related biomechanic 2b changes from baseline | Comparison at the end of the race from baseline before race
  To study the relationship between the pair of shoes worn and the morphological, biomechanical and sensory characteristics of the ultra-endurance runner- Measurement of foot dimensions (scanner)
  - Measurement of biomechanics ( stride frequency)
shoes related biomechanic 2c changes from baseline | Comparison at the end of the race from baseline before race
  To study the relationship between the pair of shoes worn and the morphological, biomechanical and sensory characteristics of the ultra-endurance runner- Measurement of foot dimensions (scanner)
  - Measurement of biomechanics (ground contact time)
shoes related biomechanic 3a changes from baseline | Comparison at the end of the race from baseline before race
  To study the relationship between the pair of shoes worn and the morphological, biomechanical and sensory characteristics of the ultra-endurance runner- Measurement of foot dimensions (scanner)
  - Collection and measurement of the characteristics of the shoes used (brand)
shoes related biomechanic 3b changes from baseline | Comparison at the end of the race from baseline before race
  To study the relationship between the pair of shoes worn and the morphological, biomechanical and sensory characteristics of the ultra-endurance runner- Measurement of foot dimensions (scanner)
  - Collection and measurement of the characteristics of the shoes used (model)
shoes related biomechanic 3c changes from baseline | Comparison at the end of the race from baseline before race
  To study the relationship between the pair of shoes worn and the morphological, biomechanical and sensory characteristics of the ultra-endurance runner- Measurement of foot dimensions (scanner)
  - Collection and measurement of the characteristics of the shoes used (size)
shoes related biomechanic 3d changes from baseline | Comparison at the end of the race from baseline before race
  To study the relationship between the pair of shoes worn and the morphological, biomechanical and sensory characteristics of the ultra-endurance runner- Measurement of foot dimensions (scanner)
  - Collection and measurement of the characteristics of the shoes used (sole thickness)
shoes related biomechanic 3e changes from baseline | Comparison at the end of the race from baseline before race
  To study the relationship between the pair of shoes worn and the morphological, biomechanical and sensory characteristics of the ultra-endurance runner- Measurement of foot dimensions (scanner)
  - Collection and measurement of the characteristics of the shoes used (drop)
shoes related biomechanic 3f changes from baseline | Comparison at the end of the race from baseline before race
  To study the relationship between the pair of shoes worn and the morphological, biomechanical and sensory characteristics of the ultra-endurance runner- Measurement of foot dimensions (scanner)
  - Collection and measurement of the characteristics of the shoes used (internal pressures)
Psychology and performances changes from baseline | pre day 1 before, per (lap 1 to 6) and post measurments day 1 after the race
  Two computerized 2D tests (money risk test described in Schmidt et al. Plos biology 2012)
glycemia regulation changes from baseline | continuous monitoring from two days before the race up to one seven day after the race
  Evaluate the impact of ultra trail on the glycemic balance of Runners through a continuous interstitial glucose sensor (FreeStyle Libre Pro, Abbott): continuous measurment of capillar glycemia
Fatigue and biomechanics 1 changes from baseline | pre day 1 before, per (lap 1 to 6) and post measurments day 1 after the race
  Study the effects of fatigue on the biomechanics of running :running kinematics, mainly the foot placement on the ground measured with high definition video camera
Fatigue and biomechanics 2 changes from baseline | pre day 1 before, per (lap 1 to 6) and post measurments day 1 after the race
  Study the effects of fatigue on the biomechanics of running :running kinematics, mainly the pace of the steps measured with an optogait system.

CONTACTS AND LOCATIONS:
Overall Officials: stephane Besnard, MD, Principal Investigator — CaenHU
Locations (1):
- Clecy Center, Clécy, France

REFERENCES:
- [Derived] Parent C, Mauvieux B, Lespagnol E, Hingrand C, Vauthier JC, Noirez P, Hurdiel R, Martinet Q, Delaunay PL, Besnard S, Heyman J, Gabel V, Baron P, Gamelin FX, Maboudou P, Rabasa-Lhoret R, Jouffroy R, Heyman E. Glycaemic Effects of a 156-km Ultra-trail Race in Athletes: An Observational Field Study. Sports Med. 2024 Aug;54(8):2169-2184. doi: 10.1007/s40279-024-02013-4. Epub 2024 Mar 30. PMID 38555307